CLINICAL TRIAL: NCT07143435
Title: Endoscopic Findings in Iron Deficiency Anemia: A Cross-Sectional Study From Port Sudan
Acronym: IDA
Status: Completed | Type: Observational
Sponsor: National Center for Gastroentestinal and Liver Disease (Other)
Responsible Party: Sponsor
Other Study IDs: EndoscopicFindingsIronDef
Record Dates: First submitted 2025-08-09; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Iron Deficiency Anemia; Endoscopy; Anemia
Keywords: Sudan; Gastrointestinal blood loss; Endoscopic findings
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Iron deficiency anemia (IDA) is a common condition often linked to gastrointestinal blood loss, making endoscopic evaluation essential for identifying underlying causes. This study aimed to assess the endoscopic findings in patients presenting with IDA in Red Sea State, Sudan. Understanding the prevalence and types of gastrointestinal lesions among these patients can aid in early diagnosis and management, reducing associated morbidity and mortality. By focusing on patients undergoing endoscopic evaluation, this study provides valuable insights into the burden of gastrointestinal pathologies contributing to IDA in the region.

Materials and Methods: This cross-sectional, descriptive study was conducted in the Endoscopy Unit at Alkaleej Medical Complex - Portsudan. Adults aged ≥18 years with IDA undergoing endoscopic evaluation were included, excluding those unwilling participation or with incomplete data. Data were collected via structured questionnaires and medical records, covering demographics, medical history, clinical presentation, and endoscopic findings. SPSS version 26 - 2018, was used for analysis, applying descriptive statistics and chi-square tests to assess associations. Ethical approval was obtained, and informed consent was secured from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above.
* Patients diagnosed with IDA who underwent endoscopic evaluation.

Exclusion Criteria:

* Patients who declined to participate in the study.
* Patients with incomplete medical records or missing endoscopic findings.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of all patients presenting with IDA who underwent endoscopic evaluation at the study site during the study period.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with endoscopic lesions explaining iron deficiency anemia | 4 months
  Percentage of participants with one or more endoscopic findings potentially accounting for IDA (e.g., gastric/duodenal ulcer, gastritis with bleeding, colonic mass/ulcer, angiodysplasia), confirmed by endoscopy ± biopsy when indicated.

SECONDARY OUTCOMES:
Proportion of biopsy-proven malignancies | 4 months
  Percentage of participants with histopathology-confirmed gastrointestinal malignancy (e.g., gastric adenocarcinoma, colorectal cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ganim, Dr., Study Director — National Center for Gastrointestinal And Liver Diseases
Locations (1):
- Alkhaleej Medical Center, Kassala, Sudan